CLINICAL TRIAL: NCT02401685
Title: POSNOC - POsitive Sentinel NOde: Adjuvant Therapy Alone Versus Adjuvant Therapy Plus Clearance or Axillary Radiotherapy. A Randomised Controlled Trial of Axillary Treatment in Women With Early Stage Breast Cancer Who Have Metastases in One or Two Sentinel Nodes
Brief Title: POSNOC - A Trial Looking at Axillary Treatment in Early Breast Cancer
Acronym: POSNOC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Collaborators: University of Nottingham (Other); Sussex Health Outcomes Research & Education in Cancer (SHORE-C) (Unknown); NCRI Radiotherapy Trials QA Group (RTTQA) (Unknown); Breast Cancer Trials, Australia and New Zealand (Other)
Responsible Party: Principal Investigator, Dr Amit Goyal, Consultant Oncoplastic Breast Surgeon & Associate Professor, University Hospitals of Derby and Burton NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RD-5103-001-13; ISRCTN Number (Registry Identifier: ISRCTN54765244)
Record Dates: First submitted 2015-03-11; First posted 2015-03-30 (Estimated); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
Keywords: breast cancer; sentinel lymph node biopsy; axillary lymph node clearance; axillary lymph node dissection; macrometastases; axillary radiotherapy; POSNOC
MeSH Terms: conditions — Breast Neoplasms | interventions — Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adjuvant therapy alone (Experimental): Women in this arm will have adjuvant therapy but no treatment to their armpit after surgery. Axillary and supraclavicular fossa radiotherapy is not allowed when randomised to this arm.
  Interventions: Other: Adjuvant therapy
- Adjuvant therapy plus axillary treatment (Active Comparator): Women in this arm will have adjuvant therapy plus treatment to their armpit after surgery. Axillary treatment can be axillary node clearance or axillary radiotherapy as per local guidelines.
  Interventions: Other: Adjuvant therapy; Procedure: Axillary treatment

INTERVENTIONS:
Other: Adjuvant therapy — Adjuvant therapy will include chemotherapy and/or endocrine therapy for all women, and radiotherapy to breast or chest wall if indicated. Human epidermal growth factor receptor 2 (HER2) targeted treatment may also be administered when indicated.
Procedure: Axillary treatment — Axillary treatment can be axillary node clearance or axillary radiotherapy as per local guidelines.
  Arms: Adjuvant therapy plus axillary treatment

SUMMARY:
POSNOC is a pragmatic, randomised, multicentre, non-inferiority trial.

Aim For women with early stage breast cancer and one or two sentinel node macrometastases, to assess whether adjuvant therapy alone is no worse than adjuvant therapy plus axillary treatment, in terms of axillary recurrence within 5 years.

Stratification: Institution, Age (<50, ≥50), Breast-conserving surgery (BCS) or mastectomy, Estrogen receptor (ER) status (positive, negative), Number of positive nodes (1, 2), Intra-operative sentinel assessment using OSNA (yes, no).

Interventions The study will compare adjuvant therapy alone with adjuvant therapy plus axillary treatment (axillary node clearance (ANC) or axillary radiotherapy (ART)).

Sample Size: 1900 participants

Follow-up: Participants will be followed up for 5 years.

Adjuvant Therapy: All participants will receive adjuvant systemic therapy (chemotherapy and/or endocrine therapy). All participants may receive breast/chest wall radiotherapy. Axillary and supraclavicular fossa radiotherapy is not allowed when randomised to adjuvant therapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Unifocal or multi-focal invasive tumour with lesion ≤5 cm in its largest dimension, measured pathologically or largest invasive tumour diameter on radiology should be used for women who are randomised intra-operatively or undergo sentinel node biopsy before neoadjuvant therapy (tumour size should be based only on the single largest tumour; do not add the sizes together from the multiple foci)
* At sentinel node biopsy have 1 or 2 nodes with macrometastases (tumour deposit >2.0mm in largest dimension or defined as macrometastasis on molecular assay)
* Fit for axillary treatment and adjuvant therapy
* Have given written informed consent

Exclusion Criteria:

* bilateral invasive breast cancer
* more than 2 nodes with macrometastases
* neoadjuvant therapy for breast cancer except:

  * if sentinel node biopsy performed prior to neoadjuvant chemotherapy in women with early breast cancer
  * short duration of neoadjuvant endocrine therapy is acceptable (up to 3 months)
* previous axillary surgery on the same body side as the scheduled sentinel node biopsy
* not receiving adjuvant systemic therapy
* previous cancer less than 5 years previously or concomitant malignancy except:

  * basal or squamous cell carcinoma of the skin
  * in situ carcinoma of the cervix
  * in situ melanoma
  * contra- or ipsilateral in situ breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1900 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Axillary recurrence | 5 years
  Axillary recurrence is defined as pathologically (cytology or biopsy) confirmed recurrence in lymph nodes draining the primary tumour site.

SECONDARY OUTCOMES:
Arm morbidity | 3 years
  Arm morbidity will be assessed by the Lymphoedema and Breast Cancer and QuickDASH (disabilities of the arm, shoulder and hand) questionnaires.
Quality of life | 3 years
  Quality of life will be assessed using the Functional Assessment of Cancer Therapy-Breast+4 questionnaire.
Anxiety (Spielberger State/Trait Anxiety Inventory) | 3 years
  Anxiety will be assessed with the Spielberger State/Trait Anxiety Inventory.
Economic evaluation (EQ-5D-5L (EuroQoL) | 3 years
  Health-related quality of life will be evaluated using the EQ-5D-5L (EuroQoL) instrument.
Local (breast or chest wall) recurrence | 5 years
  Number of participants with local (breast or chest wall) recurrence.
Regional (nodal) recurrence | 5 years
  Number of participants with regional (nodal) recurrence.
Distant metastasis | 5 years
  Number of participants with distant metastasis.
Time to axillary recurrence | 5 years
Axillary recurrence free survival | 5 years
Disease free survival | 5 years
Overall survival | 5 years
Contralateral breast cancer | 5 years
  Number of participants with contralateral breast cancer.
Non-breast malignancy | 5 years
  Number of participants with non-breast malignancy.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Goyal, Principal Investigator — University Hospitals of Derby and Burton NHS Foundation Trust
Locations (50):
- Australia (8):
  - Royal Adelaide Hospital, Adelaide
  - Bankstown-Lidcocombe Hospital, Bankstown
  - Maeter Hospital, Brisbane
  - Coffs Harbour Health Campus, Coffs Harbour
  - Monash Cancer Centre, Melbourne
  - Royal Melbourne and Royal Women's Hospital, Melbourne
  - Sir Charles Gairdner Hospital, Perth
  - Riverina Cancer Care Centre, Wagga Wagga
- New Zealand (2):
  - Waikato Hospital, Hamilton
  - Rotorua Hospital, Rotorua
- United Kingdom (40):
  - Ashford and St Peter's Hospitals NHS Foundation Trust, Ashford
  - Barnsley Hospital, Barnsley
  - Belfast City Hospital, Belfast
  - City Hospital, Birmingham
  - Queen Elizabeth Hospital, Birmingham
  - Royal Bolton Hospital, Bolton
  - Bradford Royal Infirmary, Bradford
  - Princess of Wales Hospital, Bridgend
  - Addenbrooke's Hospital, Cambridge
  - University Hospital Llandough, Cardiff
  - Darrent Valley Hospital, Dartford
  - Royal Derby Hospital, Derby
  - Eastbourne District General Hospital, Eastbourne
  - Western General Hospital, Edinburgh
  - Medway Maritime Hospital, Gillingham
  - Western Infirmary, Glasgow
  - Inverclyde Royal Hospital, Greenock
  - Harrogate District Hospital, Harrogate
  - University Hospital Crosshouse, Kilmarnock
  - Forth Valley Hospital, Larbert
  - St James's University Hospital, Leeds
  - University Hospitals of Leicester NHS Trust, Leicester
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Royal Marsden Hospital, London
  - Luton and Dunstable University Hospital, Luton
  - Macclesfield District General Hospital, Macclesfield
  - Maidstone Hospital, Maidstone
  - North Manchester General Hospital, Manchester
  - Wythenshawe Hospital, Manchester
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Royal Gwent Hospital, Newport
  - The Norfolk and Norwich University Hospital, Norwich
  - Oxford University Hospitals, Oxford
  - Peterborough City Hospital, Peterborough
  - Derriford Hospital, Plymouth
  - Rotherham General Hospital, Rotherham
  - Royal Stoke University Hospital, Stoke-on-Trent
  - Royal Cornwall Hospital, Truro
  - Wishaw General Hospital, Wishaw
  - New Cross Hospital, Wolverhampton

REFERENCES:
- [Background] Goyal A, Dodwell D. POSNOC: A Randomised Trial Looking at Axillary Treatment in Women with One or Two Sentinel Nodes with Macrometastases. Clin Oncol (R Coll Radiol). 2015 Dec;27(12):692-5. doi: 10.1016/j.clon.2015.07.005. Epub 2015 Aug 5. No abstract available. PMID 26254841
- [Background] Dodwell D, Goyal A. Axillary conservation in early breast cancer. Br J Surg. 2015 Oct;102(11):1297-9. doi: 10.1002/bjs.9881. Epub 2015 Jul 7. No abstract available. PMID 26148870
- [Background] Goyal A, Dodwell D, Reed MW, Coleman RE. Axillary treatment in women with one or two sentinel nodes with macrometastases: more evidence is needed to inform practice. J Clin Oncol. 2014 Dec 1;32(34):3902. doi: 10.1200/JCO.2014.57.3717. Epub 2014 Sep 22. No abstract available. PMID 25245444
- See also: Trial website — http://www.posnoc.co.uk
- See also: X/twitter account — https://x.com/posnoc